CLINICAL TRIAL: NCT04043143
Title: 24-hour Oral Morphine Equivalent Based Opioid Prescribing After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18-2098; K23DA040923 (NIH)
Record Dates: First submitted 2019-04-18; First posted 2019-08-02 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Opioid Use
Keywords: opioids

STUDY DESIGN:
Intervention Model Description: The investigators will test this tool prospectively for Cesarean section patients anticipated to use about half or less of the usually prescribed amount of opioid pain pills randomized equally to prescription tool intervention or no intervention (prescription as usual).
Who Masked: Participant, Investigator
Masking Description: The investigators will use an electronic randomization scheme created so that the principal investigator and statistician can remain blind to assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Prescription As Usual (Placebo Comparator): At the time of writing the discharge prescription for a patient the provider will receive a best practice alert (BPA) to consider prescribing the usual medications for pain management after discharge.
  Interventions: Other: Arm 1 Prescription As Usual
- Arm 2 Prescription Tool Intervention (Experimental): At the time of writing the discharge prescription for a patient the provider will be informed by the best practice alert (BPA) Prescription Tool that a patient may be considered for a lower post-discharge opioid dose (no opioids for patients who did not take any opioids in the last 24 hours, and 10 oxycodone 5mg tablets, for patients having taken less than 22.5 MME, e.g. 1-3 oxycodone 5mg tablets in the last 24 hours). Final dosing decisions and drug choices will remain at the discretion of the treating provider and decisions will be tracked.
  Interventions: Other: Arm 2 Prescription Tool Intervention

INTERVENTIONS:
Other: Arm 1 Prescription As Usual — At the time of writing the discharge prescription for a patient the provider will receive a best practice alert (BPA) to consider prescribing the usual medications for pain management after discharge.
  Arms: Arm 1 Prescription As Usual
Other: Arm 2 Prescription Tool Intervention — The best practice alert (BPA) Prescription Tool will only make a suggestion to the provider if the patient may be considered for a lower post-discharge opioid dose. Providers may still choose to prescribe a higher dose as clinically indicated.
  Arms: Arm 2 Prescription Tool Intervention

SUMMARY:
The investigators will utilize the electronic health record to individualize pain therapy in surgical patients after hospital discharge using last 24-hour opioid intake as the decision variable for the amount of opioid pain pills prescribed. The preliminary data indicate that current opioid prescription practice after surgery follows a "one size fits all" pattern. In-hospital opioid use 24 hours prior to discharge serves as a strong indicator to correctly estimate needs for analgesic medications at home. The investigators will test the hypothesis that this prescription estimation tool will enable providers to write need-based prescriptions based on each patient's' 24-hour prior-to-discharge opioid use. The investigators will test this tool prospectively for patients after Cesarean section who are anticipated to use about half or less of the usually prescribed amount of opioid pain pills after discharge randomized equally to prescription tool intervention or no intervention (prescription as usual).

DETAILED DESCRIPTION:
Prescription opioid overdose has emerged as a leading cause of death in the general population. Opioid-based therapy represents a corner-stone of post-operative pain management. With increasing emphasis on robust pain therapy, sales of opioid medications have increased four-fold in the last decade. Parallel to this rise, opioid-associated deaths have also quadrupled. The investigators have shown that long-term opioid use occurs in up to 22% of patients following surgery. Over-prescribed opioids after surgery can create a reservoir of opioids that become available for non-medical use. Effective strategies to maximize non-opioid pain therapy and to limit such a reservoir are lacking. Thus, there is an urgent need to individualize post-operative pain therapy and reduce reliance on opioids.

Converting knowledge on actual need for opioid pain medications after surgery into tangible benefits can prevent over-prescription of opioids that become available for non-medical use. The objective of this study is to prescribe pain medications after surgery in a patient-centered fashion. The investigators will use the average amount of opioid medications (in oral morphine equivalents - OME) taken in the last 24 hours prior to discharge to inform and design a clinical decision support tool. This tool will reduce the amount of opioid medications prescribed while maintaining patient post-operative pain control. The calculated "last 24 hour OME dose" will be applied to generate a recommendation for the prescription of a cumulative opioid dose that will be shared with the provider when the post-discharge pain medication is made, e.g. via displaying the last 24-hour opioid use in the electronic health record (EHR). The rationale is that testing of such a decision-making tool will lay the groundwork to translate the findings of this project into more secure and efficient opioid prescribing practices to a system-wide level. Upon completion, the investigators expect to have developed an effective decision-making tool to help providers estimate required pain medication following patient discharge.

The investigators will perform a randomized clinical trial (RCT) of an Electronic Health Record (EHR)-based recommendation to prescribe opioids at discharge according to the recorded last 24-hour inpatient use according to current recommendations and evaluate its effect on the amount of opioids prescribed as well as pain control after discharge.

Using the University of Colorado Hospital Epic/Clarity database, the investigators will continuously identify all patients who underwent Cesarean section surgery at University Hospital. Patients will be approached regarding interest in the study prior to hospital discharge.A trained Professional Research Assistant or other provider will explain the study and obtain informed consent from prospective participants. After consent, demographics and the best contact information will be collected from those enrolled patients who indicate they are interested in completing the surveys after their hospital discharge.

The investigators expect 44 patients to complete all four weekly surveys and define the intent-to-treat sample as patients who complete one or more surveys (providing at least one observation to be used in analyses). To conservatively allow for increased variability due to attrition, 54 patients will be randomized equally electronically to intervention (prescription tool) or no intervention (prescription as usual). The investigators will use an electronic randomization scheme created so that the principal investigator and statistician can remain blind to assignment.

In the intervention group (Arm 2), at the time of writing the prescription for a patient, the provider will be informed that a patient may be considered for a lower post-discharge opioid dose (No opioids for patients who did not take any opioids in the last 24 hours, and 10 oxycodone 5mg tablets, for patients having taken equal or less than 22.5 MME (morphine milligram equivalent), e.g. 1-3 oxycodone 5mg tablets in the last 24 hours.) In the control group (Arm 1), providers will receive a message to consider prescribing the usual medications for pain management after discharge. Final dosing decisions and drug choices will remain at the discretion of the treating provider and decisions will be tracked. For this pilot study, the provider information (best practice alert - BPA) will be operationalized via a written recommendation on paper handed to the provider by study staff in a sealed envelope that the provider will be asked to open and read. Alternatively the BPA may be presented electronically using a screen. Providers will be asked to acknowledge that they read the BPA by closing the window or opening the envelope.

One week after hospital discharge interested patients will be contacted and asked to complete the first of four surveys. All communication will be available in English. Patients will be paid with a $10 gift card or money order equivalent to complete the study assessments using REDCap at each of the four weekly follow-up time points ($40 total). All enrolled patients will complete the weekly post-discharge surveys within REDCap or hard copy if they do not have internet access.

The study team will contact all subjects ~2 weeks after discharge to ask about pain management and monitor the need for secondary prescriptions from providers to ensure that no significant under-prescription of opioid medications after surgery occurs.

The investigators will seek follow-up with providers about the usefulness and acceptability of the EHR-based intervention. Providers will be surveyed with a REDCap survey using a modified version of the GUIDES checklist, which provides a tool to improve the successful use of guideline-based computerized clinical decision support.

ELIGIBILITY:
Inclusion Criteria:

* Women ages at least 18 years of age having undergone Cesarean section surgery at the University of Colorado Hospital are eligible.
* Willingness to complete weekly surveys for 4 weeks after discharge.
* Anticipated to need half or less of the usually prescribed amount of opioids based on the amount of opioids taken in the last 24 hours prior to the opioid medication being written for discharge (only patients who took 22.5 MME or less opioids in the last 24 hours prior to the day of discharge will be eligible for this study).

Exclusion Criteria:

* Patients under the age of 18 years.
* Patients returning to institutional settings (e.g. prison, jail, mental health facility).
* Pregnant women (patients will be approached after their C-section).
* Decisionally challenged patients.
* Blind or illiterate patients.

Based on prior research factors such as emergency status, prior opioid use, repeat vs primary C-section, and associated procedures were not associated with post-discharge opioid use once the investigators adjusted for last-24 hour inpatient opioid use. Hence, these patients will not be excluded.

Inclusion and exclusion criteria (including the amount of opioids taken in the last 24 hours prior to discharge) will be evaluated in the morning in patients scheduled to be discharged later that day.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data may be shared with other researchers as required by some journals or as requested by qualified investigators as determined by the study PI. However, all names and any other information that identifies research subjects will always be kept confidential and will not be shared.

REFERENCES:
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Background] Chen EY, Marcantonio A, Tornetta P 3rd. Correlation Between 24-Hour Predischarge Opioid Use and Amount of Opioids Prescribed at Hospital Discharge. JAMA Surg. 2018 Feb 21;153(2):e174859. doi: 10.1001/jamasurg.2017.4859. Epub 2018 Feb 21. PMID 29238810
- [Background] Volkow ND, Frieden TR, Hyde PS, Cha SS. Medication-assisted therapies--tackling the opioid-overdose epidemic. N Engl J Med. 2014 May 29;370(22):2063-6. doi: 10.1056/NEJMp1402780. Epub 2014 Apr 23. No abstract available. PMID 24758595
- [Background] Bartels K, Fernandez-Bustamante A, McWilliams SK, Hopfer CJ, Mikulich-Gilbertson SK. Long-term opioid use after inpatient surgery - A retrospective cohort study. Drug Alcohol Depend. 2018 Jun 1;187:61-65. doi: 10.1016/j.drugalcdep.2018.02.013. Epub 2018 Mar 27. PMID 29627407
- [Background] Bartels K, Binswanger IA, Hopfer CJ. Sources of Prescription Opioids for Nonmedical Use. J Addict Med. 2016 Mar-Apr;10(2):134. doi: 10.1097/ADM.0000000000000192. No abstract available. PMID 26985647
- [Background] Hill MV, Stucke RS, Billmeier SE, Kelly JL, Barth RJ Jr. Guideline for Discharge Opioid Prescriptions after Inpatient General Surgical Procedures. J Am Coll Surg. 2018 Jun;226(6):996-1003. doi: 10.1016/j.jamcollsurg.2017.10.012. Epub 2017 Nov 30. PMID 29198638
- [Background] National Institutes of Health, PROMIS tools for pain intensity and pain interference. http://www.healthmeasures.net/explore-measurement-systems/promis Last accessed on 03/02/2018.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew prior to being randomized.
Period: Overall Study
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Started | 29 | 27
Completed | 23 | 22
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 5 | 5
Not completed — screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics data is only available for the participants who completed the study (i.e. had at least one survey completed).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Prescribed Post-discharge Opioids
Description: Prescribed post-discharge opioid doses in oral morphine equivalents from the electronic health record (EHR).
Time Frame: Date of admission to the hospital up to 60 days after the date of hospital discharge.
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalent units (OME)
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 22
Oral Morphine Equivalent units (OME) | 55.3 (37.1) | 62.8 (32.8)

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 1
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 1 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: One week after hospital discharge date.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 22
T-Score Metric | 62.0 (6.4) | 58.0 (9.6)

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 2
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 2 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Two weeks after hospital discharge date.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 22
T-Score Metric | 55.2 (9.1) | 51.9 (8.2)

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 3
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 3 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Three weeks after hospital discharge date.
Population: 2 participants in Arm 2 did not complete the survey.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 20
T-Score Metric | 50.1 (8.1) | 48.6 (8.8)

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 4
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 4 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Four weeks after hospital discharge date.
Population: One participant from Arm 1 and two participants from Arm 2 did not complete the survey.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 22 | 20
T-Score Metric | 47.4 (6.9) | 46.3 (8.5)

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 1
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 1 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: One week after hospital discharge date.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 22
T-Score Metric | 58.3 (6.4) | 55.6 (8.1)

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 2
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 2 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Two weeks after hospital discharge date.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 22
T-Score Metric | 53.3 (6.5) | 49.9 (8.0)

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 3
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 3 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Three weeks after hospital discharge date.
Population: 2 participants in Arm 2 did not complete the survey.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 23 | 20
T-Score Metric | 48.6 (6.3) | 45.2 (8.5)

9. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 4
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 4 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Four weeks after hospital discharge date.
Population: One participant from Arm 1 and two participants from Arm 2 did not complete the survey.
Measure: Mean (Standard Error); unit: T-Score Metric
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
Number analyzed (Participants) | 22 | 20
T-Score Metric | 45.2 (6.1) | 43.6 (9.2)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: Only participants who completed the study (i.e. completed at least one survey after discharge) were analyzed for adverse events.
Arm/Group | Arm 1 Prescription As Usual | Arm 2 Prescription Tool Intervention
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT04043143/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT04043143/ICF_001.pdf